CLINICAL TRIAL: NCT03330327
Title: An Open Label, Fixed-Sequence, Glucose Clamp Study to Compare Molar Potency of HM12470 and Regular Human Insulin in Healthy Subjects
Brief Title: Molar Potency Study of HM12470 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HM-INS-115-102
Record Dates: First submitted 2017-10-26; First posted 2017-11-06 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1 (Experimental): Intravenous (IV) infusion of HM12470
  Interventions: Biological: HM12470
- Part 2: Sequence 1 (Experimental): Intravenous (IV) infusion of HM12470
  Interventions: Biological: HM12470
- Part 2: Sequence 2 (Experimental): Intravenous (IV) infusion of HM12470
  Interventions: Biological: HM12470

INTERVENTIONS:
Biological: HM12470 — HM12470 is a long-acting insulin analogue

SUMMARY:
This is a phase 1 study to assess and compare molar potency of HM12470 and regular human insulin in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Females must be non-pregnant and non-lactating
* Males must be surgically sterile or using an acceptable contraceptive method

Exclusion Criteria:

* Participation in an investigational study within 30 days prior to dosing
* Use of new prescription and non-prescription drugs within 3 weeks preceding the first dosing

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2015-03-30 (Actual); Primary Completion 2017-08-17 (Actual); Study Completion 2017-08-17 (Actual)

PRIMARY OUTCOMES:
Blood glucose assessment of HM12470 and regular human insulin (RHI) over the entire dosing period | 1 month
  - Comparison of HM12470 to RHI based on blood glucose profile generated by intravenous infusion

SECONDARY OUTCOMES:
Cmax of HM12470 | 1 month
  - Maximum concentration of HM12470 over the entire dosing period
AUC of HM12470 | 1 month
  - Area Under the Curve of HM12470 over the entire dosing period

CONTACTS AND LOCATIONS:
Locations (1):
- Hanmi Investigative Site, Chula Vista, California, United States

IPD SHARING:
Plan to Share IPD: Undecided